CLINICAL TRIAL: NCT04837313
Title: Efficacy and Safety of Fecal Microbiota Transplantation in the Treatment of Parkinson's Disease With Constipation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou First People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K-2020-107-02
Record Dates: First submitted 2020-12-20; First posted 2021-04-08 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2020-10

CONDITIONS: Parkinson's Disease; Fecal Microbiota Transplantation
MeSH Terms: conditions — Parkinson Disease | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parkinson's Disease with Constipation (Experimental): Fecal microbiota transplantation will be performed.
  Interventions: Procedure: Fecal Microbiota Transplantation

INTERVENTIONS:
Procedure: Fecal Microbiota Transplantation — Fecal Microbiota Transplantation

SUMMARY:
Parkinson's disease(PD) may cause the autonomic nervous system's improper functioning, which is responsible for regulating the intestinal tract movement. A certain degree of degeneration of digestive system function can cause PD patients to constipation symptoms. Studies have shown that up to 63 percent of people with Parkinson's disease experience constipation. What is more, medications for PD, including levodopa and dopamine agonist, can also cause constipation. In recent years, an increasing number of studies have been conducted to investigate gut microflora and their influence on the central nervous system. Furthermore, some studies of Parkinson's disease have confirmed that gut microflora plays a vital role in the occurrence and development of Parkinson's disease.

The purpose of this study is to evaluate the efficacy and safety of fecal microbiota transplantation in the treatment of constipation symptoms in patients with Parkinson's disease receiving a steady dose of levodopa. We will also analyze intestinal flora diversity in patients with Parkinson's disease with constipation. The investigation of the gut microbiome may emerge as a new therapeutic measure to treat constipation associate with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-75 years of age
* Signed informed consent form
* Clinical diagnosis of Parkinson's disease (according to 2016 edition of Chinese Parkinson's disease diagnostic criteria)
* Parkinson's disease duration of 1 year or more
* Hoehn & Yahr stage 1-4 (including)
* Patients have following 2 or more symptoms, which appear for at least 6 months and exist in recent 3 months: A. at least 25% of defecation feel strenuous; B. At least 25% of defecation was not massive or hard; C. at least 25% of defecation had incomplete feeling; D. at least 25% of defecation had anorectal obstruction; E. at least 25% of defecation needed manual assistance; F. defecation less than 3 times a week, with or without abdominal pain
* Patients are taking oral L-dopa (with or without Benserazide, carbidopa, and O-methyltransferase inhibitors) at least 4 weeks, and be able to tolerate a steady dose of dopamine agonists, monoamine oxidase B inhibitors, anticholinergics, and / or adamantine.
* Patients are taking stable dosage of anti-PD drugs, antidepressant drugs and antipsychotics for more than 1 month.
* Be able to tolerate the FMT infusion method such as endoscopy, colonoscopy, capsule, nasoduodenal tube insertion, etc.
* Be able to receive follow-up visit, follow-up examination and specimen collection on time

Exclusion Criteria:

* Patients with Parkinson's syndrome and Parkinsonism plus syndrome
* History of cerebrovascular accident, brain injury, epilepsy and other brain injury
* The "opening" stage was Hoehn & Yahr 5
* Patient received neurosurgical intervention or stereotactic brain surgery for Parkinson's disease
* Patients with organic lesions of digestive tract
* Patients had major abdominal surgery
* History of infectious diarrhea and took antibiotics in recent 2 weeks
* Patients infected with Clostridium difficile and other pathogens
* Patients with HIV or compromised immune system (such as congenital immunodeficiency or currently taking immunosuppressive drugs)
* Patients with uncontrollable basic diseases of digestive system
* Patients could not fully understand and sign the informed consent form
* Patients who were not considered suitable for inclusion in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The Efficacy of FMT in patients with constipation will be assessed by the change of The Gastrointestinal Symptom Rating Scale (GSRS) and Wexner Constipation Score. | 6 months
  The data will be collected in several time points from baseline to 6 months after FMT. Gastrointestinal Symptom Rating Scale(GSRS) is a measure of gastrointestinal symptom severity in five clusters (pain, bloating, constipation, diarrhea, and early satiety).The items are scored between 1 and 7, where 1 corresponds to "no discomfort at all" and 7 to "very severe discomfort" from the symptom.
  Wexner Constipation Scoring system is a scale to evaluate the severity of constipation. These factors included frequency of bowel movements, painful evacuation, incomplete evacuation, abdominal pain, length of time per attempt, assistance for evacuation, unsuccessful attempts for evacuation per 24 hours, and duration of constipation, with 0 indicating normal and 30 indicating severe constipation.

SECONDARY OUTCOMES:
The improvement of clinical symptoms in patients with Parkinson's Disease will be assessed by the change of several scales of Parkinson's Disease. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hongli Huang, MM, Principal Investigator — Guangzhou First People's Hospital
Locations (1):
- Guangzhou First People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baizabal-Carvallo JF. Gut microbiota: a potential therapeutic target for Parkinson's disease. Neural Regen Res. 2021 Feb;16(2):287-288. doi: 10.4103/1673-5374.290896. No abstract available. PMID 32859778
- [Background] Bhattarai Y, Kashyap PC. Parkinson's disease: Are gut microbes involved? Am J Physiol Gastrointest Liver Physiol. 2020 Nov 1;319(5):G529-G540. doi: 10.1152/ajpgi.00058.2020. Epub 2020 Sep 2. PMID 32877215
- [Background] Dutta SK, Verma S, Jain V, Surapaneni BK, Vinayek R, Phillips L, Nair PP. Parkinson's Disease: The Emerging Role of Gut Dysbiosis, Antibiotics, Probiotics, and Fecal Microbiota Transplantation. J Neurogastroenterol Motil. 2019 Jul 1;25(3):363-376. doi: 10.5056/jnm19044. PMID 31327219
- [Background] Mhyre TR, Boyd JT, Hamill RW, Maguire-Zeiss KA. Parkinson's disease. Subcell Biochem. 2012;65:389-455. doi: 10.1007/978-94-007-5416-4_16. PMID 23225012
- [Background] Yang D, Zhao D, Ali Shah SZ, Wu W, Lai M, Zhang X, Li J, Guan Z, Zhao H, Li W, Gao H, Zhou X, Yang L. The Role of the Gut Microbiota in the Pathogenesis of Parkinson's Disease. Front Neurol. 2019 Nov 6;10:1155. doi: 10.3389/fneur.2019.01155. eCollection 2019. PMID 31781020
- [Background] Stocchi F, Torti M. Constipation in Parkinson's Disease. Int Rev Neurobiol. 2017;134:811-826. doi: 10.1016/bs.irn.2017.06.003. Epub 2017 Jul 13. PMID 28805584